CLINICAL TRIAL: NCT04286165
Title: A Randomized Controlled Trial Comparing Brief Peer Supported webSTAIR to Enhanced Wait List
Brief Title: Brief Peer Supported webSTAIR Compared to Enhanced Wait List
Acronym: BPSwS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Responsible Party: Principal Investigator, Marylène Cloitre, Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CLO0009
Record Dates: First submitted 2020-01-08; First posted 2020-02-26 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Post Traumatic Stress Disorder; Depression; Emotion Regulation
Keywords: PTSD; Post Traumatic Stress Disorder; Depression; Emotion Regulation; Skills Building; Peer; Coaching; Online
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression; Emotional Regulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BPS webSTAIR 6 Levels with Peer Support (Active Comparator): Participants in BPS webSTAIR will complete a baseline, posttreatment and 2-month follow-up assessment. In the BPS webSTAIR condition, participants will first complete a welcome module to orient them to the program. After randomization, participants will have 10 weeks to complete the 6 modules. Every time the Veteran logs on they will have the opportunity to engage with a Veteran peer for support through the web program. Contacts can last for up to an hour. Veterans will receive a series of automated reminders and engagement emails that the Vets Prevail program sends at various points in the program.
  Interventions: Other: Brief Peer Supported webSTAIR
- Wait List (No Intervention): In Wait list, participants will be asked to go about their life as usual. They will be asked not to participate in any other programs for PTSD or depression symptoms for 10 weeks. After the 10 weeks, WL participants can begin any other program for PTSD or depression. They will also be given the option of participating in BPS webSTAIR or be provided with information about other web-based programs that might be of interest or relevant to them.

INTERVENTIONS:
Other: Brief Peer Supported webSTAIR — The BPS webSTAIR program is an online platform where individuals are taught skills in emotion regulation. In this program they will learn how to recognize the emotions they are feeling by assessing their own body language, being attentive to their thought processes, and attempting to replace negative behaviors with positive. Throughout the platform they will engage in written exercises to help them solidify the lessons with their own life experiencing. They will also have the support of peers throughout the program to help them when they need clarification or having a difficult time applying the lesson(s).
  Arms: BPS webSTAIR 6 Levels with Peer Support

SUMMARY:
This study will enroll 180 Veterans at a 2:1 ratio where 120 Veterans will be enrolled into a brief transdiagnostic peer supported webSTAIR (BPS webSTAIR) and 60 will be supported into Waitlist. The purpose of the study is to assess the efficacy BPS webSTAIR in regard to four outcomes: reduction in PTSD and depression symptoms (measured by the PCL-5 and PHQ-8, respectively) and improvement in emotion regulation and work and social adjustment (measured by the DERS-16 and WSAS, respectively). The active treatment is a 6-session modular treatment that focuses on learning emotion management skills where Particpants will have 10 weeks to complete the treatment. Assessments will occur three times for those in webSTAIR: baseline, post-treatment (10 weeks after randomization) and 8-week follow-up and twice for those on waitlist (baseline and 10 weeks after randomization). It is hypothesized that BPS WebSTAIR will be superior to the Waitlist condition on all four outcomes. Mixed Effects Models will be used to evaluate the outcomes.

DETAILED DESCRIPTION:
The purpose of this randomized controlled trial is to assess the efficacy of a brief version of webSTAIR (BPS webSTAIR) supported by peers compared to a waitlist condition (WL). Brief peer supported (BPS) webSTAIR is a 6-module web-based transdiagnostic program that provides skills training in emotion regulation; participants in this condition will be able to contact a Veteran peer trained in the program to obtain general support plus guidance about program use and application of skills.

An 11-module version of webSTAIR with therapist coaching has provided pilot data that the program is effective in reducing symptoms of posttraumatic stress disorder (PTSD) and depression as well as improving emotion regulation and work and social adjustment. Pilot data indicate that initial gains are made in the first 6 sessions. In addition, qualitative interviews with Veterans who have completed the program indicate high satisfaction with these modules. This study will assess whether a shorter version of the treatment (6 rather than 11 modules) and with peer rather than professional coaching will be effective compared to a waitlist condition. The BPS webSTAIR program was developed with the aim of providing a treatment for trauma-related symptoms that is effective, brief, engaging and likely to be completed by the user. The reduction of the number of modules creates a briefer treatment than the investigators current web-based program. In addition, data indicated that integrating Veteran peers into mental health programs leads to better engagement and greater retention providing the rationale for including Veteran peers rather than therapists (e.g., psychologists, social workers). Given the absence of findings that a brief, peer-supported version of webSTAIR provides improvement in the above symptoms, the research team followed recommendations for the development and testing of psychotherapies and used a waitlist control as an initial test of efficacy.

The aim is to establish the efficacy of BPS webSTAIR in improving symptoms of PTSD and depression, emotion regulation problems and work and social adjustment compared to a Waitlist Control.

Hypothesis 1a: Compared to WL, BPS webSTAIR will provide greater improvement in PTSD symptoms as measured by the PCL5 and depression as measured by the PHQ-8 (secondary outcome). Assessments will be made at pre-treatment, post-treatment, and 8-week follow-up for webSTAIR participants and pre and post-treatment (or 10 weeks from randomization) for WL.

Hypothesis 1b: Compared to WL, BPS webSTAIR will provide greater improvement in emotion regulation as measured by the DERS-16 and overall functioning as measured by the work and social adjustment scale (WSAS) (secondary outcomes). Assessments will be made at pre-treatment, post-treatment and 8-week follow-up for webSTAIR participants and pre and post-treatment (or 10 weeks after randomization) for WL.

In the BPS webSTAIR condition, participants will first complete a welcome module to orient them to the program. After randomization, participants will have 10 weeks to complete the 6 modules. Every time the Veteran logs on they will have the opportunity to engage with a Veteran peer for support through the web program. Contacts can last for up to an hour. Veterans will receive a series of automated reminders and engagement emails that the Vets Prevail program sends at various points in the program.

The equivalence of the treatment conditions on baseline variables demographics and psychological variables) will be assessed and controlled (if necessary) in the final analyses. Other preliminary analyses will include examination of distributional properties of the measures. Transformations will be used to improve distributions when necessary. Missing data patterns (from missed assessments and from dropout) will be examined and compared between conditions. Mixed Effects Models (MEMs) will be used to evaluate differences between the two treatments over time with time as a main effect and treatment-by-time as an interaction term.

ELIGIBILITY:
Inclusion Criteria:

* Able to read/write English
* Internet connection allowing stable access to VetsPrevail website
* Have experienced at least one traumatic event (positive on the LEC)
* A score greater than or equal to 3 on the PC-PTSD OR greater than or equal to 2 on the PHQ2 on the screen.
* Enrollment into the webSTAIR study must be completed within two weeks of completing screener/eligibility based on symptoms.

Exclusion Criteria:

* Currently receiving a trauma-focused intervention (PE, CPT, EMDR, WET) assessed during baseline
* Being unlikely to benefit from therapy or Telemental health, for example:
* Cognitive difficulties as indicated during baseline assessment.
* Active psychosis as indicated during baseline assessment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Change from Baseline on PTSD Checklist for DSM-5 (PCL-5) at program completion and at two months after program completion. | Before the participant is randomized. 10 weeks from randomization. 2 months after the participant finishes all 6 levels of the intervention for participants engaged in treatment.
  The PTSD Checklist for DSM-5 (PCL-5) is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The PCL-5 has a variety of purposes, including, monitoring symptom change during and after treatment, screening individuals for PTSD and making a provisional PTSD diagnosis. The scale ranges from Not At All (0) to Extremely (4) Higher scores relate to more severe symptoms.
Change from Baseline on Personal Health Questionnaire Depression Scale (PHQ - 8) at program completion and at two months after program completion. | Before the participant is randomized. 10 weeks from randomization. 2 months after the participant finishes all 6 levels of the intervention for participants engaged in treatment.
  The eight-item Personal Health Questionnaire Depression Scale (PHQ - 8) is established as a valid diagnostic and severity measure for depressive disorders in large clinical studies.The scale ranges from Not At All (1) to Nearly Every Day (4) Higher scores relate to more severe symptoms.
Change from Baseline on Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) at program completion and at two months after program completion. | Before the participant is randomized. 10 weeks from randomization. 2 months after the participant finishes all 6 levels of the intervention for participants engaged in treatment.
  Difficulties in Emotion Regulation Scale - 16 item version (DERS-16) is a widely-used, theoretically-driven, and psychometrically-sound self-report measure of emotion regulation difficulties. The scale ranges from Almost Never (1) to Almost Always (5). Higher scores relate to more severe symptoms.
Change from Baseline on The Work and Social Adjustment Scale (WSAS) at program completion and at two months after program completion. | Before the participant is randomized. 10 weeks from randomization. 2 months after the participant finishes all 6 levels of the intervention for participants engaged in treatment.
  The The Work and Social Adjustment Scale (WSAS) is a measure of people's problems sometimes affect their ability to do certain day-to-day tasks in their lives. To rate your problems, look at each section and determine on the scale provided how much your problem impairs your ability to carry out the activity in the past month.The scale ranges from No Impairment (0) to Very Severe Impairment (8). Higher scores relate to more severe impairment.
Life Events Checklist for DSM-5 (LEC-2) | Before the participant is randomized to a condition.
  The Life Events Checklist for DSM-5 (LEC-2) lists difficult or stressful things that sometimes happen to people. Mark the item for any single stressful event you have experienced. Be sure to consider your entire life (growing up, as well as adulthood) as you go through the list of events. You do not need to answer any of these questions if doing so would be distressing. The scale consists of Yes, No and Prefer Not To Answer. More Yes responses indicate experiencing more traumatic events in a participant's history.

CONTACTS AND LOCATIONS:
Overall Officials: Marylene Cloitre, PhD, Principal Investigator — National Center for PTSD Dissemination and Training Division
Locations (1):
- VA Palo Alto Health Care System, NC-PTSD, Dissemination and Training Division, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ong LE, Speicher S, Villasenor D, Kim J, Jacobs A, Macia KS, Cloitre M. Brief Peer-Supported Web-Based Skills Training in Affective and Interpersonal Regulation (BPS webSTAIR) for Trauma-Exposed Veterans in the Community: Randomized Controlled Trial. J Med Internet Res. 2024 Oct 2;26:e52130. doi: 10.2196/52130. PMID 39012722

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT04286165/Prot_SAP_000.pdf